CLINICAL TRIAL: NCT03201770
Title: Phase IIIb/IV Cohort Event Monitoring Study To Evaluate, In Real Life Setting, The Safety And Tolerability In Malaria Patients Of The Fixed-Dose Artemisinin-Based Combination Therapy Pyramax®
Brief Title: Cohort Event Monitoring Study of Pyramax®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-021-15
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2018-01

CONDITIONS: Malaria,Falciparum
Keywords: Uncomplicated Malaria; Pyramax; Pyronaridine artesunate
MeSH Terms: conditions — Malaria, Falciparum | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyramax (Experimental): Pyronaridine artesunate tablets (180/60mg) and granules (60/20mg)
  Interventions: Drug: pyronaridine artesunate

INTERVENTIONS:
Drug: pyronaridine artesunate — Antimalarial treatment
  Other Names: Pyramax

SUMMARY:
The study is to be performed in public health facilities in Central and West Africa where Pyramax will be used as treatment of uncomplicated malaria episodes, including repeat episodes. The study is to assess the safety of Pyramax, particularly in patients with underlying liver function abnormalities, in patients who have co-morbid conditions, such as HIV, and also in very small children (<1 year of age).

DETAILED DESCRIPTION:
This is a non-comparative Cohort Event Monitoring study. The study will assess the safety of Pyramax in terms of the evaluation and identification of the hepatic safety events in a sub group of patients enrolled with liver function tests (LFT)s >2x upper limit of normal (ULN) from blood taken immediately prior to treatment without any clinical signs or symptoms of hepatotoxicity and with signs and symptoms of uncomplicated malaria confirmed by a Rapid Diagnostic Test (RDT) or microscopy (thick blood smear). The study will compare the clinical hepatic safety of Pyramax between a cohort of patients enrolled with LFTs >2xULN and a cohort of patients enrolled with normal LFTs matched for demographic characteristics.

An estimated 8,572 malaria episodes are to be recruited to provide 120 malaria episodes in patients with baseline raised LFTs >2xULN for follow up of liver function. A cohort of at least 2% of children who are <1 year of age will be included for monitoring of liver function.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated malaria (Plasmodia of any species) diagnosed as per national policies and in line with WHO recommendations:

  * Fever or history of fever in the previous 24 h and/or the presence of anaemia, for which pallor of the palms appears to be the most reliable sign in young children.
  * Confirmation of malaria by a parasitological diagnosis (RDT or Microscopy (thick blood smear). analysis).
* Weight ≥5 kg - < 20 kg (granules); ≥20 kg (tablets).
* Ability to take an oral medication.
* Ability and willingness to participate based on signed informed consent (a parent or a guardian has to sign for children below 18 years old) and on signed assent form for minors that could be required per national regulations in each participating country.
* The patient has to comply with all scheduled follow-up visits.

Exclusion Criteria:

* Patients with clinical signs or symptoms of hepatic injury (such as nausea, abdominal pain associated with jaundice) or known severe liver disease (i.e. decompensated cirrhosis, Child-Pugh stage 3 or 4).
* Known allergy to artemisinin and/or to pyronaridine.
* Known pregnancy.
* Lactating women should be excluded if other anti-malarial treatments are available.
* Complicated malaria as per WHO definition (Annex 2)
* Patients that the investigator considers would be at particular risk if receiving an anti-malarial or if participating in the study.
* Patients having been treated with Pyramax in the previous 28 days.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8572 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Evaluation and identification of hepatic safety events, including raised liver function tests | Assessment up to Day 28.
  Evaluation and identification of hepatic safety events (including raised liver function tests - LFTs) of Pyramax in a sub group of malaria patients enrolled with LFTs >2xUL.

SECONDARY OUTCOMES:
Overall safety | Assessment up to Day 28.
  Evaluation of the adverse event reporting of Pyramax in the treatment of uncomplicated malaria under real life conditions.
Evaluation of Efficacy | Assessment up to Day 28.
  Evaluation of the efficacy based on crude Day 28 cure rate by species and PCR adjusted cure rate for Day 28 cure rate for P. falciparum of Pyramax in the treatment of uncomplicated malaria under real life conditions

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramharter, MD, DTM&H, Principal Investigator — CERMEL, University of Tübingen, Germany
Locations (5):
- The Biotechnology Center Nkolbisson, Univ of Yaounde I, Messa, Yaoundé, Cameroon
- Institut Pierre Richet / Institut National de SanPublique (IPR/INSP), Bouaké, Côte d’Ivoire
- Centre de Recherche du Centre Hospitalier du Mont Amba, Kinshasa, Democratic Republic of the Congo
- CERMEL, Albert Schweitzer Hospital, Lambaréné, Gabon
- Centre de Santé FCRM, Hospital of Talangai, Brazzaville, Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramharter M, Djimde AA, Borghini-Fuhrer I, Miller R, Shin J, Aspinall A, Richardson N, Wibberg M, Fleckenstein L, Arbe-Barnes S, Duparc S. Safety and efficacy of pyronaridine-artesunate paediatric granules in the treatment of uncomplicated malaria in children: insights from randomized clinical trials and a real-world study. Malar J. 2024 Feb 28;23(1):61. doi: 10.1186/s12936-024-04885-3. PMID 38418982
- [Derived] Koehne E, Zander N, Rodi M, Held J, Hoffmann W, Zoleko-Manego R, Ramharter M, Mombo-Ngoma G, Kremsner PG, Kreidenweiss A. Evidence for in vitro and in vivo activity of the antimalarial pyronaridine against Schistosoma. PLoS Negl Trop Dis. 2021 Jun 24;15(6):e0009511. doi: 10.1371/journal.pntd.0009511. eCollection 2021 Jun. PMID 34166393
- [Derived] Tona Lutete G, Mombo-Ngoma G, Assi SB, Bigoga JD, Koukouikila-Koussounda F, Ntamabyaliro NY, Ntoumi F, Agnandji ST, Groger M, Shin J, Borghini-Fuhrer I, Arbe-Barnes S, Allen SJ, Kremsner PG, Miller R, Duparc S, Ramharter M; CANTAM study group. Pyronaridine-artesunate real-world safety, tolerability, and effectiveness in malaria patients in 5 African countries: A single-arm, open-label, cohort event monitoring study. PLoS Med. 2021 Jun 15;18(6):e1003669. doi: 10.1371/journal.pmed.1003669. eCollection 2021 Jun. PMID 34129601